CLINICAL TRIAL: NCT05544396
Title: Study on the Probiotics Regulating miRNA in H. Pylori-induced Wnt/β-catenin Gastric Carcinogenesis.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yao-Jong Yang, professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-106-085
Record Dates: First submitted 2022-07-06; First posted 2022-09-16 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: H. Pylori Infection; Carcinogenesis
Keywords: H. Pylori; Wnt/beta-catenin; miRNA; carcinogenesis
MeSH Terms: conditions — Carcinogenesis | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic group (Experimental): Routine eradicate treatment H. pylori, and probiotics (2 packs per day) for 6 months.
  Interventions: Other: probiotic
- control group (Placebo Comparator): Only routine eradicate treatment H. pylori.
  Interventions: Other: probiotic

INTERVENTIONS:
Other: probiotic — probiotic group give probiotics (2 packs per day) for 6 months.

SUMMARY:
Background. H. pylori has recognized as a type 1 carcinogen for gastric adenocarcinoma. Although H. pylori eradication promises to reduce the risk of gastric cancer, the regression rate of intestinal metaplasia (IM) after eradication is unsatisfactory. Therefore, to find the mechanism of IM persistent and a new strategy to improve IM regression are critical for reducing gastric cancer development. The canonical Wnt/beta-catenin signaling pathway upregulating cyclooxygenase-2 (COX-2) transcriptional activity involves gastric carcinogenesis after H. pylori infection. Investigators have established an in vitro model that H. pylori induces a cagA-dependent nuclear COX-2 expression in both GES-1 and AGS cells. MicroRNAs (miRNAs) are a class of widespread non-coding RNAs and have been shown to involve in the gastric carcinogenesis. Among these gastric cancer-related miRNA candidates, some were reported to interact with Wnt/β-catenin pathway. Clinically, H. pylori eradication plus celecoxib therapy results in about one-third cases being IM regression, which correlated to the nuclear β-catenin and COX-2 expression before treatment. Based on the probiotics ingestion can ameliorate H. pylori-induced inflammatory pathways, investigators hypothesis that H. pylori eradication with probiotics supplement may promote IM regression through regulating certain miRNAs and Wnt/β-catenin signaling. The aims of this 3-year grant will

1. to establish the H. pylori induces the Wnt/beta-catenin and COX-2 signaling pathway in vitro.
2. to investigate the effects and mechanisms of L. acidophilus and B. latis on H. pylori-induced Wnt/beta-catenin oncogenesis pathway.
3. to study whether probiotics ingestion promote IM regression or ameliorate IM progression in H. pylori-infected patients after successful eradication therapy.

Materials and Methods. A H. pylori (HP238) isolate strain, GES-1, and AGS cells will be used for in vitro study. The protein levels of cell tests will measured by western blot. The differences of miRNAs expression between monk, cells infected with H. pylori, and cells pretreated with probiotics than infected by H. pylori will be analyzed by next generation sequencing method. H. pylori-infected patients with IM will be randomly allocated to receive probiotics or controls, the 2nd endoscopy will be arranged at the 12th month to evaluate the IM status.

Anticipated results. This study will to establish the H. pylori-induced Wnt/beta-catenin oncogenesis pathway in vitro. Furthermore, the effect and mechanism of probiotics inhibit the H. pylori-induced Wnt/beta-catenin signaling will be clarified. Finally, investigators will provide an evidence for the probiotics ingestion promote the rate of IM regression in patients after H. pylori eradication.

DETAILED DESCRIPTION:
What are already know

1. H. pylori-induced Wnt/beta-catenin cascades leads to gastric carcinogenesis.
2. Nuclear beta-catenin and COX-2 expression correlated to the IM regression rate in human after H. pylori eradication.
3. Administration of selective COX-2 inhibitos, celecoxib, results in partial IM regression in patients with long-term IM persistence after H. pylori eradication
4. Certain miRNAs involve in gastric oncogenesis by targeting Wnt/beta-catenin signaling pathway.

What will be add

1. The Wnt/beta-catenin oncogenesis induction is different between primary (GES-1), and cancer (AGS) gastric cells after H. pylori infection.
2. Probiotics ameliorate or prevent H. pylori-induced gastric Wnt/beta-catenin/COX2 carcinogenesis signaling through regulating miRNAs.
3. Probiotics administration improves regression rate in patients with CAG and IM after H. pylori successful eradication.

Diagram of clinical trial to evaluate probiotics ingestion improves H. pylori-related intestinal metaplasia (IM) in patients after eradication therapy

A.The dyspeptic patients receiving PES and biopsies will be continuously enrolled to find H. pylori infection and IM.

B.Investigators keep to allocate patients into probiotics-treatment and controls (each group 30 patients).

C.To compare the miRNA(s) serum levels in patients with IM regression and IM persistent by real-time PCR.

D.To analyze the significance of probiotics ingestion improves IM regression rate in the RTC.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* Have undergone gastroscopy
* First discovered H.pylori infection and intestinal metaplasia

Exclusion Criteria:

* Massive bleeding is life-threatening
* Gastric cancer
* Previous treatment for H.pylori
* Long-term use of non-steroidal anti-inflammatory drugs (eg, aspirin), and hydrogen ion pump inhibitors.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
The IM regression rate one year after H. pylori eradication | Eligible participants allocated to treat or non-treat groups. The panendoscopy was performed one year later.
  H. pylori-infected participants (n=100) with IM received successful H. pylori eradication.
  Group I (n=50) given oral probiotics 1 pack bid for 6 months, Group II did not treat.
  The 2nd panendoscopy followed at one year later to evaluate IM status using Updated Sydney System Score.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University & Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The whole IPD will be shared after 2026.

REFERENCES:
- [Background] Sheu BS, Tsai YC, Wu CT, Chang WL, Cheng HC, Yang HB. Long-term celecoxib can prevent the progression of persistent gastric intestinal metaplasia After H. pylori eradication. Helicobacter. 2013 Apr;18(2):117-23. doi: 10.1111/hel.12013. Epub 2012 Sep 26. PMID 23067366
- [Background] Hung KH, Wu JJ, Yang HB, Su LJ, Sheu BS. Host Wnt/beta-catenin pathway triggered by Helicobacter pylori correlates with regression of gastric intestinal metaplasia after H. pylori eradication. J Med Microbiol. 2009 May;58(Pt 5):567-576. doi: 10.1099/jmm.0.007310-0. PMID 19369517
- [Derived] Yang YJ, Wu CT, Cheng HC, Chen WY, Tseng JT, Chang WL, Sheu BS. Probiotics ameliorate H. pylori-associated gastric beta-catenin and COX-2 carcinogenesis signaling by regulating miR-185. J Biomed Sci. 2025 Jun 3;32(1):55. doi: 10.1186/s12929-025-01149-3. PMID 40462044